CLINICAL TRIAL: NCT00320606
Title: Immunosuppression Withdrawal for Pediatric Living-donor Liver Transplant Recipients (ITN029ST)
Brief Title: Withdrawal of Immunosuppression in Pediatric Liver Transplant Recipients
Acronym: WISP-R
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN029ST
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Liver Transplant; Liver Transplantation
Keywords: immunosuppression withdrawal (IS); anti-rejection drugs; tolerance; allograft function

STUDY DESIGN:
Intervention Model Description: Recipients of parental living-donor liver allografts will undergo gradual withdrawal as tolerated of immunosuppression with the goal of complete withdrawal.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immunosuppression Withdrawal (Experimental): Recipients of parental living donor liver transplants 4 or more years prior to trial enrollment, who also had stable allograft function during the preceding 6 months while taking a single immunosuppressive drug were permitted to undergo withdrawal of immunosuppression therapy. With high dose, daily dose reduction by 25% for 8 weeks. With low dose, daily dose reduction by 25% for 4 weeks.
  Participants are carefully evaluated/monitored throughout the study by assessments including but not limited to liver biopsy, liver tests and clinic visits, alloantibodies, autoantibodies and quantitative immunoglobulin G test results.
  Interventions: Drug: Immunosuppression Withdrawal

INTERVENTIONS:
Drug: Immunosuppression Withdrawal — Gradual withdrawal of immunosuppressive medication. With high dose, daily dose reduction by 25% for 8 weeks. With low dose, daily dose reduction by 25% for 4 weeks.
  Other Names: ISW

SUMMARY:
Antirejection medicines, also known as immunosuppressive drugs, are prescribed to organ transplant recipients to prevent their bodies from rejecting the new organ. Long-term use of these drugs places transplant recipients at higher risk of serious infections and certain types of cancer. The purpose of this study is to determine whether immunosuppressive drugs can be safely withdrawn over a minimum of 9 months from children who received liver transplants at least 4 years ago.

DETAILED DESCRIPTION:
In order to prevent the rejection of transplanted organs, transplant recipients are prescribed a strict, lifelong regimen of immunosuppressive drugs. While these drugs help prevent the body from rejecting the transplant, they carry numerous complications, including increased risk of serious infections and certain types of cancer. However, there is mounting evidence that a significant percentage of liver transplant recipients can maintain a healthy, functioning transplant without ongoing immunosuppression. This study will determine whether gradual withdrawal and eventual discontinuation of all immunosuppressive medication can be safely accomplished in children who received a liver transplant from a parent. Twenty eligible participants who were under 18 years old at the time of transplant, whose donor was a parent, and who received the transplant at least four years ago will be enrolled in the study.

Liver recipients will have an initial screening assessment consisting of a medical history, liver biopsy, and urine and blood collection. Eligible recipients will be placed on a modified medication schedule to gradually decrease their immunosuppression medication slowly over a 9- to 12-month period, during which time they will be closely monitored by study staff. Immunosuppressive drugs will not be provided by this study. For a minimum of 3 and up to a maximum of 7 years, monthly telephone consultations and quarterly study visits will occur. Visits will include physical exams and blood collection to monitor the children's health during the withdrawal phase. The exact schedule of immunosuppressant withdrawal will be determined by study physicians based on participant's health and immune function test results. Donor and nondonor parents will be asked to each provide one blood sample during the initial study visits for immunologic and genetic testing.

*** IMPORTANT NOTICE: *** The National Institute of Allergy and Infectious Diseases and the Immune Tolerance Network do not recommend the discontinuation of immunosuppressive therapy for recipients of cell, organ, or tissue transplants outside of physician-directed, controlled clinical studies. Discontinuation of prescribed immunosuppressive therapy can result in serious health consequences and should only be performed in certain rare circumstances, upon the recommendation and with the guidance of your health care provider.

ELIGIBILITY:
Inclusion Criteria for Liver Recipients:

* Received liver from living parent donor
* Received transplant at least 4 years prior to study entry
* Less than 18 years of age at time of transplant
* Parent or guardian willing to provide informed consent

Inclusion Criteria for Liver Donors:

* Willing to participate in this study

Exclusion Criteria for Liver Recipients:

* Underwent transplant because of liver failure related to autoimmune disease
* Underwent transplant of a second organ simultaneously with or after liver transplant OR liver retransplantation
* Receiving immunosuppression with more than one drug
* 50% increase in dose of current immunosuppressive drug
* HIV infection
* Hepatitis B or C virus infection
* Pregnancy or breastfeeding

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06-05 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Feng, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional study materials are available to the public in: 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from Division of Allergy, Immunology, and Transplantation (DAIT)-funded grants and contracts and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal.
Time Frame: Already available to the public.
Access Criteria: Available to the public. Study ID is SDY662:WISP-R ITN029ST
URL: http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY662

REFERENCES:
- [Background] Reding R. Long-term complications of immunosuppression in pediatric liver recipients. Acta Gastroenterol Belg. 2005 Oct-Dec;68(4):453-6. PMID 16433002
- [Result] Feng S, Ekong UD, Lobritto SJ, Demetris AJ, Roberts JP, Rosenthal P, Alonso EM, Philogene MC, Ikle D, Poole KM, Bridges ND, Turka LA, Tchao NK. Complete immunosuppression withdrawal and subsequent allograft function among pediatric recipients of parental living donor liver transplants. JAMA. 2012 Jan 18;307(3):283-93. doi: 10.1001/jama.2011.2014. PMID 22253395
- [Result] Perito ER, Mohammad S, Rosenthal P, Alonso EM, Ekong UD, Lobritto SJ, Feng S. Posttransplant metabolic syndrome in the withdrawal of immunosuppression in Pediatric Liver Transplant Recipients (WISP-R) pilot trial. Am J Transplant. 2015 Mar;15(3):779-85. doi: 10.1111/ajt.13024. Epub 2015 Feb 3. PMID 25648649
- [Result] Feng S, Demetris AJ, Spain KM, Kanaparthi S, Burrell BE, Ekong UD, Alonso EM, Rosenthal P, Turka LA, Ikle D, Tchao NK. Five-year histological and serological follow-up of operationally tolerant pediatric liver transplant recipients enrolled in WISP-R. Hepatology. 2017 Feb;65(2):647-660. doi: 10.1002/hep.28681. Epub 2016 Jul 27. PMID 27302659
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network website — https://www.immunetolerance.org/
- Available data/document: Individual Participant Data Set: SDY662:WISP-R ITN029ST — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY662 — ImmPort study identifier is Study ID is SDY662:WISP-R ITN029ST
- Available data/document: Study summary, -schematic, -detailed description, -download packages et al.: SDY662:WISP-R ITN029ST — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY662 — ImmPort study identifier is Study ID is SDY662:WISP-R ITN029ST
- Available data/document: Individual Participant Data Set: WISP-R ITN029ST — http://www.itntrialshare.org/project/Studies/ITN029STJAMA/Study%20Data/begin.view — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available without charge. Creating an account for ITN TrialShare is free and allows for searching studies of interest.
- Available data/document: Study protocol synopsis, -navigator, abstracts and manuscripts, datasets et al.: WISP-R ITN029ST — https://www.itntrialshare.org/project/Studies/ITN029STJAMA/Study%20Data/begin.view — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available without charge. Creating an account for ITN TrialShare is free and allows for searching studies of interest.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three centers in the United States enrolled 20 pediatric recipients of parental living-donor liver allografts between June 2006 and August 2008.
Pre-assignment Details: Informed consent was obtained from eligible individuals prior to screening assessments. Participants then underwent procedures at screening to determine eligibility according to the study's inclusion/exclusion criteria.
Groups:
- Immunosuppression Withdrawal Arm: Participants were gradually tapered off of their single immunosuppression (IS) drug (cyclosporine or tacrolimus), over a 36 week period by first reducing the drug dose and then the dosing frequency until the participant was completely withdrawn from all immunosuppression.
Period: Overall Study
Arm/Group | Immunosuppression Withdrawal Arm
Started | 20
Completed | 17
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.7 (2.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Baseline Glomerular Filtration Rate (GFR) [Median (Inter-Quartile Range); unit: mL/min/1.73 m^2] — Glomerular filtration rate (GFR) is a measure of kidney function. The bedside Schwartz equation was used to estimate GFR from serum creatinine and height in children. Baseline serum creatinine was utilized in this equation, defined as the creatinine value at the start of immunosuppressive (IS) treatment tapering. Baseline height was utilized in the equation, defined as the last height recorded prior to the start of IS treatment tapering. Estimate of normal GFR: ≥90 mL/min per 1.73 m^2.
  mL/min/1.73 m^2 | 113.2 [93.40 to 121.13]
Baseline Total Cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Total serum cholesterol collected at the start of IS tapering.
  Target range for total cholesterol: 75-169 mg/dL if age ≤20; high values indicate risk of cardiovascular disease
  mg/dL | 147 [132 to 162]
Baseline Glucose [Median (Inter-Quartile Range); unit: mg/dL] — Glucose collected at the start of tapering. This is a measure of glucose found in the blood. Glucose, a sugar, is an energy source that the body relies on to properly function. If levels are too high for a long period of time, diabetes can develop. Diabetes can result in many long-term complications such as eye, kidney, and nerve damage, stroke, and cardiovascular complications.
  Target range for fasting glucose: 60-106 mg/dL.
  mg/dL | 89.5 [84.0 to 94.0]
Baseline Systolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] — Systolic blood pressure measured at the start of IS tapering. Systolic blood pressure measures the pressure on the blood vessels when the heart beats and thus is pushing blood to the rest of the body. For pediatric participants, normal systolic blood pressure is defined as being below the 90th percentile for the participant's age, sex, and height on at least 3 separate occasions. High blood pressure, also known as hypertension, is a risk factor for coronary artery disease, stroke, heart failure, and other complications if left unmanaged.
  mmHg | 109.5 [100.0 to 117.5]
Baseline Diastolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] — Diastolic blood pressure measured at the start of IS tapering. Diastolic blood pressure measures the pressure in the arteries when the heart is a rest and is thus filled with blood. For pediatric participants, normal systolic blood pressure is defined as being below the 90th percentile for the participant's age, sex, and height on at least 3 separate occasions. High blood pressure, also known as hypertension, is a risk factor for coronary artery disease, stroke, heart failure, and other complications if left unmanaged.
  mmHg | 64.5 [58.0 to 73.5]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Successfully Withdrawn From Immunosuppression
Description: Participants were considered successfully withdrawn from immunosuppression if they remained off immunosuppression for at least one year with normal allograft function.
Time Frame: 1 year after completion of immunosuppression withdrawal
Population: Intent-to-Treat
Measure: Number; unit: Proportion of participants
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 20
Proportion of participants | 0.60
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal Arm; The proportion of participants in whom immunosuppression withdrawal was attempted who are successfully withdrawn from immunosuppression are descriptively summarized with 95% confidence intervals using an exact binomial method; Test type: Other; 95% confidence interval using an exact b = 0.6, 95% CI 2-sided [0.4 to 0.8] — Proportion Success

2. Secondary Outcome: Number of Participants Who Suffered Graft Loss or Died Following Initiation of Immunosuppression Withdrawal
Description: Participants who died while on the study for any reason as well as participants that experienced the loss of their transplant while a participant in the study.
Time Frame: Enrollment through end of study (up to 9.5 years)
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 20
Participants | 0
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal Arm; The proportion of participants in whom immunosuppression (IS) withdrawal was attempted who are successfully withdrawn from immunosuppression and experience death or graft loss are descriptively summarized with 95% confidence intervals using an exact binomial method; Test type: Other; Binomial Proportion = 0, 95% CI 2-sided [0.0 to 0.1684] — 95% Confidence Interval Exact Binomial

3. Secondary Outcome: Time From Start of Immunosuppression Withdrawal to the First Episode of Acute Rejection, Second Episode of Rejection That Did Not Require Treatment, or to Diagnosis of Chronic Rejection
Description: The number of days between the start of immunosuppression (IS) withdrawal and the first episode of acute rejection (either clinical rejection or based on BANFF criteria), second episode of rejection that did not require treatment, or the first diagnosis of chronic rejection.
Time Frame: From the start of immunosuppression withdrawal to first acute rejection, second episode of rejection that did not require treatment, or diagnosis of chronic rejection through end of study (up to 9.5 years)
Population: Intent-to-Treat participants who experienced acute rejection or were diagnosed with chronic rejection.
Measure: Mean (95% Confidence Interval); unit: Days
Groups:
- Immunosuppression Withdrawal Arm: Participants were gradually tapered off of their single immunosuppression drug (cyclosporine or tacrolimus), over a 36 week period by first reducing the drug dose and then the dosing frequency until the participant was completely withdrawn from all immunosuppression.
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 7
Days | 211.57 [113.56 to 309.58]

4. Secondary Outcome: Immunosuppression-Free Duration
Description: The number of months between the end of immunosuppression withdrawal and either the end of trial participation or the time of restarting immunosuppression
Time Frame: Completion of Withdrawal to either end of trial participation (up to 9.5 years) or time to restarting immunosuppression
Population: Intent-to-Treat participants who completed withdrawal
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 15
Months | 75.84 [53.28 to 98.39]

5. Secondary Outcome: Distribution of Histologic Severity Among Rejection Episodes
Description: The number of participants within each level of histologic severity based on BANFF grading criteria (Mild, Moderate, Severe).
Time Frame: Start of immunosuppressive withdrawal to rejection through end of study (up to 9.5 years)
Population: Participants from the Intent-to-treat group who experienced a biopsy-proven rejection episode
Measure: Number; unit: Biopsy Proven rejection episodes
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 4
Biopsy Proven rejection episodes
  Mild | 3
  Moderate | 2
  Severe | 0

6. Secondary Outcome: Number of Participants Experiencing Adverse Events by Severity
Description: The results provide the total number of participants experiencing adverse events (AEs). Participants experiencing AEs are stratified into five severity categories: mild, moderate, severe, life-threatening, and death, based on National Cancer Institute--Common Terminology Criteria (NCI-CTCAE) Version 3.0.
Time Frame: Enrollment through end of study (up to 9.5 years)
Population: Intent-To-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 20
Participants
  Total Adverse Events | 19
  Mild | 18
  Moderate | 17
  Severe | 6
  Life Threatening | 0
  Death | 0

7. Secondary Outcome: Percent Change From Baseline in Renal Function Measured by the Glomerular Filtration Rate (GFR)
Description: Percent change from baseline at each annual visit. The bedside Schwartz equation was used to estimate GFR from serum creatinine and height in children. Baseline serum creatinine was utilized in the equation, defined as the creatinine value at the start of IS tapering. Baseline height was utilized in the equation, defined as the last height recorded prior to the start of IS tapering. Serum creatinine measurements and height measurements at the annual visits were used to calculate the annual GFR. When height value was not available, the height collected prior to the annual visit was used in the GFR calculation. M12 and M24 visits represent Medium Frequency visits; L12 and L24 represent low frequency visits, and E12-48 represent extended follow-up visits.
Time Frame: Enrollment through end of study (up to 9.5 years)
Population: Intent-To-Treat with GFR data at visits available for analysis
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 18
Percent change
  Percent Change in GFR at Month 12: number analyzed (Participants) | 9
  Percent Change in GFR at Month 12 | 4.5 [2.41 to 22.42]
  Percent Change in GFR at M12 Visit | 8.7 [3.89 to 28.05]
  Percent Change in GFR at M24 Visit: number analyzed (Participants) | 12
  Percent Change in GFR at M24 Visit | 20.5 [5.46 to 48.40]
  Percent Change in GFR at L12 Visit: number analyzed (Participants) | 12
  Percent Change in GFR at L12 Visit | 10.8 [-1.71 to 34.89]
  Percent Change in GFR at L24 Visit: number analyzed (Participants) | 11
  Percent Change in GFR at L24 Visit | 7.3 [-7.86 to 38.84]
  Percent Change in GFR at E12 Visit: number analyzed (Participants) | 11
  Percent Change in GFR at E12 Visit | -3.9 [-9.97 to 31.52]
  Percent Change in GFR at E24 Visit: number analyzed (Participants) | 11
  Percent Change in GFR at E24 Visit | -6.3 [-22.18 to 23.66]
  Percent Change in GFR at E36 Visit: number analyzed (Participants) | 11
  Percent Change in GFR at E36 Visit | -5.1 [-15.76 to 15.20]
  Percent Change in GFR at E48 Visit: number analyzed (Participants) | 11
  Percent Change in GFR at E48 Visit | -15.1 [-23.38 to 2.13]

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol
Description: Percent change from baseline in total serum cholesterol. Cholesterol is a waxy substance your body needs to build cells, but too much can be a problem since it can build-up in arteries. Narrowed arteries can result in heart attack or stroke. This outcome looks at the percent change from baseline (cholesterol level at the start of IS tapering) to each annual visit. M12 and M24 visits represent Medium Frequency visits; L12 and L24 represent low frequency visits, and E12-48 represent extended follow-up visits.
Time Frame: Enrollment through end of study (up to 9.5 years)
Population: Intent-To-Treat with cholesterol data available at visit
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 13
Percent change
  Percent Change in Cholesterol at Month 12: number analyzed (Participants) | 6
  Percent Change in Cholesterol at Month 12 | -7.9 [-16.23 to -5.33]
  Percent Change in Cholesterol at M12 Visit | -0.6 [-9.74 to 4.07]
  Percent Change in Cholesterol at M24 Visit: number analyzed (Participants) | 10
  Percent Change in Cholesterol at M24 Visit | -10.9 [-14.21 to -5.92]
  Percent Change in Cholesterol at L12 Visit: number analyzed (Participants) | 11
  Percent Change in Cholesterol at L12 Visit | -3.0 [-16.67 to 1.26]
  Percent Change in Cholesterol at L24 Visit: number analyzed (Participants) | 10
  Percent Change in Cholesterol at L24 Visit | -10.7 [-18.37 to -7.10]
  Percent Change in Cholesterol at E12 Visit: number analyzed (Participants) | 10
  Percent Change in Cholesterol at E12 Visit | -9.0 [-15.38 to 0.94]
  Percent Change in Cholesterol at E24 Visit: number analyzed (Participants) | 9
  Percent Change in Cholesterol at E24 Visit | -11.2 [-15.38 to -5.66]
  Percent Change in Cholesterol at E36 Visit: number analyzed (Participants) | 8
  Percent Change in Cholesterol at E36 Visit | -6.9 [-19.00 to 6.78]
  Percent Change in Cholesterol at E48 Visit: number analyzed (Participants) | 8
  Percent Change in Cholesterol at E48 Visit | -10.9 [-14.51 to 10.36]

9. Secondary Outcome: Percent Change From Baseline in Blood Glucose
Description: Glucose, a sugar, is an energy source that the body relies on to properly function. If levels are too high for a long period of time, diabetes can develop. Diabetes can result in many long-term complications such as eye, kidney, and nerve damage, stroke, and cardiovascular complications. The outcome looks at the percent change from baseline (glucose level at the start of tapering) to each annual visit. M12 and M24 visits represent Medium Frequency visits; L12 and L24 represent low frequency visits, and E12-48 represent extended follow-up visits.
Time Frame: Enrollment through end of study (up to 9.5 years)
Population: Intent-To-Treat with glucose data available at visit
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 17
Percent change
  Percent Change in Glucose at Month 12: number analyzed (Participants) | 9
  Percent Change in Glucose at Month 12 | -2.2 [-4.44 to 10.87]
  Percent Change in Glucose at M12 Visit | 1.0 [-6.32 to 13.41]
  Percent Change in Glucose at M24 Visit: number analyzed (Participants) | 12
  Percent Change in Glucose at M24 Visit | 1.8 [-5.47 to 9.41]
  Percent Change in Glucose at L12 Visit: number analyzed (Participants) | 12
  Percent Change in Glucose at L12 Visit | -0.5 [-5.42 to 9.09]
  Percent Change in Glucose at L24 Visit: number analyzed (Participants) | 11
  Percent Change in Glucose at L24 Visit | 2.0 [0.00 to 15.22]
  Percent Change in Glucose at E12 Visit: number analyzed (Participants) | 11
  Percent Change in Glucose at E12 Visit | -3.3 [-7.53 to 8.99]
  Percent Change in Glucose at E24 Visit: number analyzed (Participants) | 11
  Percent Change in Glucose at E24 Visit | -1.1 [-6.45 to 4.82]
  Percent Change in Glucose at E36 Visit: number analyzed (Participants) | 11
  Percent Change in Glucose at E36 Visit | 5.6 [-5.32 to 13.98]
  Percent Change in Glucose at E48 Visit: number analyzed (Participants) | 11
  Percent Change in Glucose at E48 Visit | -5.3 [-10.64 to 4.49]

10. Secondary Outcome: Percent Change From Baseline in Systolic Blood Pressure
Description: Systolic blood pressure (BP) measures the pressure on the blood vessels when the heart is beats and thus is pushing blood to the rest of the body. This outcome assesses the percent change from baseline (systolic blood pressure measurement at the start of tapering) to each annual visit. M12 and M24 visits represent Medium Frequency visits; L12 and L24 represent low frequency visits, and E12-48 represent extended follow-up visits.
Time Frame: Enrollment through end of study (up to 9.5 years)
Population: Intent-to-treat with systolic blood pressure data available at visit
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 17
Percent change
  Percent Change in Systolic BP at Month 12: number analyzed (Participants) | 10
  Percent Change in Systolic BP at Month 12 | 2.0 [-9.65 to 6.32]
  Percent Change in Systolic BP at M12 Visit | 0.0 [-9.65 to 5.83]
  Percent Change in Systolic BP at M24: number analyzed (Participants) | 12
  Percent Change in Systolic BP at M24 | 4.3 [-2.87 to 10.66]
  Percent Change in Systolic BP at L12 Visit: number analyzed (Participants) | 12
  Percent Change in Systolic BP at L12 Visit | 3.8 [-5.05 to 10.08]
  Percent Change in Systolic BP at L24 Visit: number analyzed (Participants) | 11
  Percent Change in Systolic BP at L24 Visit | 8.6 [2.68 to 20.41]
  Percent Change in Systolic BP at E12 Visit: number analyzed (Participants) | 11
  Percent Change in Systolic BP at E12 Visit | 2.8 [-4.46 to 14.53]
  Percent Change in Systolic BP at E24 Visit: number analyzed (Participants) | 11
  Percent Change in Systolic BP at E24 Visit | 5.1 [-3.23 to 11.67]
  Percent Change in Systolic BP at E36 Visit: number analyzed (Participants) | 11
  Percent Change in Systolic BP at E36 Visit | 9.2 [0.92 to 12.82]
  Percent Change in Systolic BP at E48 Visit: number analyzed (Participants) | 11
  Percent Change in Systolic BP at E48 Visit | 2.7 [-4.17 to 13.76]

11. Secondary Outcome: Percent Change From Baseline in Diastolic Blood Pressure
Description: Diastolic blood pressure (BP) measures the pressure in the arteries when the heart is a rest and is thus filled with blood. This outcome assesses the percent change from baseline (diastolic blood pressure measurement at the start of IS tapering) to each annual visit. M12 and M24 visits represent Medium Frequency visits; L12 and L24 represent low frequency visits, and E12-48 represent extended follow-up visits.
Time Frame: Enrollment through end of study (up to 9.5 years)
Population: Intent-to-treat with diastolic blood pressure data available at visit
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Immunosuppression Withdrawal Arm
Number analyzed (Participants) | 17
Percent change
  Percent Change in Diastolic BP at Month 12: number analyzed (Participants) | 10
  Percent Change in Diastolic BP at Month 12 | -7.5 [-15.38 to 7.41]
  Percent Change in Diastolic BP atM12 Visit | 0.0 [-8.22 to 2.70]
  Percent Change in Diastolic BP at M24 Visit: number analyzed (Participants) | 12
  Percent Change in Diastolic BP at M24 Visit | -5.4 [-16.41 to 11.92]
  Percent Change in Diastolic BP at L12 Visit: number analyzed (Participants) | 12
  Percent Change in Diastolic BP at L12 Visit | 1.5 [-12.41 to 4.73]
  Percent Change in Diastolic BP at L24 Visit: number analyzed (Participants) | 11
  Percent Change in Diastolic BP at L24 Visit | 6.6 [-9.59 to 7.59]
  Percent Change in Diastolic BP at E12 Visit: number analyzed (Participants) | 11
  Percent Change in Diastolic BP at E12 Visit | 0.0 [-7.14 to 6.06]
  Percent Change in Diastolic BP at E24 Visit: number analyzed (Participants) | 11
  Percent Change in Diastolic BP at E24 Visit | 2.6 [-5.33 to 4.55]
  Percent Change in Diastolic BP at E36 Visit: number analyzed (Participants) | 11
  Percent Change in Diastolic BP at E36 Visit | -1.4 [-8.22 to 6.58]
  Percent Change in Diastolic BP at E48: number analyzed (Participants) | 11
  Percent Change in Diastolic BP at E48 | 9.1 [-7.89 to 11.11]

ADVERSE EVENTS:
Time Frame: Enrollment through end of study (up to 9.5 years)
Description: Total number of participants in the Immunosuppression (IS) Withdrawal Arm experiencing adverse events. Participants experiencing adverse events are broken down into five severity categories, mild, moderate, severe, life-threatening, and death based on National Cancer Institute--Common Terminology Criteria (NCI-CTCAE) Version 3.0.
Arm/Group | Immunosuppression Withdrawal Arm
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 13/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunosuppression Withdrawal Arm (N=20)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (3)
Bile duct stenosis (Hepatobiliary disorders) | 3 (5)
Cholangitis (Hepatobiliary disorders) | 1 (2)
Cholangitis acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Portal vein stenosis (Hepatobiliary disorders) | 1 (1)
Transplant rejection (Immune system disorders) | 5 (5)
Enterococcal bacteraemia (Infections and infestations) | 1 (1)
Gastritis viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1)
Liver function test abnormal (Investigations) | 3 (3)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ventricular septal defect repair (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunosuppression Withdrawal Arm (N=20)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (4)
Influenza like illness (General disorders) | 9 (35)
Pyrexia (General disorders) | 4 (5)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (3)
Immunisation reaction (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (3)
Ear infection (Infections and infestations) | 3 (3)
Fungal skin infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (3)
Nasopharyngitis (Infections and infestations) | 2 (5)
Oral herpes (Infections and infestations) | 1 (1)
Pertussis (Infections and infestations) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 6 (9)
Streptococcal infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2)
Varicella (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (3)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Graft dysfunction (Injury, poisoning and procedural complications) | 1 (2)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (3)
Blood magnesium decreased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 3 (3)
Hepatic enzyme increased (Investigations) | 5 (10)
Liver function test abnormal (Investigations) | 1 (1)
Smooth muscle antibody positive (Investigations) | 1 (1)
Spleen palpable (Investigations) | 1 (1)
Vitamin D decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Growing pains (Musculoskeletal and connective tissue disorders) | 1 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Migraine (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2)
Scrotal varicose veins (Reproductive system and breast disorders) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2011-04-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT00320606/Prot_000.pdf
  • Statistical Analysis Plan (2010-04-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT00320606/SAP_001.pdf